CLINICAL TRIAL: NCT06637254
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Efficacy and Safety of HSK31858 Tablets in Patients with Bronchial Asthma
Brief Title: A Study to Evaluate the Efficacy and Safety of HSK31858 Tablets in Patients with Bronchial Asthma
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK31858-203
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-10

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HSK31858 20mg (Experimental): multiple oral doses: 20mg/d for 48w
  Interventions: Drug: HSK31858
- HSK31858 40mg (Experimental): multiple oral doses: 40mg/d for 48w
  Interventions: Drug: HSK31858
- placebo (Placebo Comparator): multiple oral doses for 48w
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK31858 — HSK31858 is a novel inhibitor of DPP1 developed by Hisco Pharmaceutical and can reduce pulmonary exacerbations over a 48-week treatment period in patients with bronchial asthma
  Arms: HSK31858 20mg; HSK31858 40mg
Drug: Placebo — the placebo comparator of study
  Arms: placebo

SUMMARY:
This is a phase II, randomised, double-blind, placebo-controlled, multicenter study to assess the efficacy and safety of HSK31858 in patients with bronchial asthma

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form.
2. Male or female patients aged ≥18 and ≤75 years at screening, weighing ≥40 kg.
3. Diagnosis of typical asthma and their history of asthma is ≥12 months at screening (provide a traceable record of asthma diagnosis).
4. Have been treated for ≥3 consecutive months prior to screening with a moderate-to-high daily dose of inhaled corticosteroids (ICS) in combination with at least one other asthma-controlling medication, and have remained stable for ≥1 month prior to screening.
5. Have had ≥1 acute exacerbation of asthma in the 12 months prior to screening.
6. Screening period (V1) pre-bronchodilator FEV1 <80% of predicted value.
7. Screening period (V1) 5-item Asthma Control Questionnaire (ACQ-5) ≥ 1.5.
8. Screening period (V1) blood eosinophil count <150/μL.
9. Female subjects with fertility or male subjects whose partner is a female with fertility must agree to have no plans to have children and to use contraception voluntarily from the time of signing the informed consent form until 3 months after the last dose. All females of childbearing potential must have a negative screening pregnancy test.
10. Subjects are able to communicate well with the investigator and are able to complete the study in accordance with the protocol requirements.

Exclusion Criteria:

1. Requires long-term oral corticosteroid maintenance therapy.
2. Subjects also have other lung diseases, including chronic obstructive pulmonary disease, bronchiectasis, and pulmonary fibrosis, not dominated by asthma as determined by the investigator.
3. Comorbid with other diseases that are clinically significant and may affect lung function, including but not limited to pleural disease, mediastinal disease, diaphragmatic lesions, myasthenia, and thoracic deformities.
4. History of malignancy: subjects with basal cell carcinoma, limited squamous cell carcinoma of the skin, or cervical carcinoma in situ will be allowed to enter the study if curative treatment has been completed for at least 12 months prior to signing the informed consent form; subjects with other malignancies will be allowed to enter the study if curative treatment has been completed for at least 5 years prior to signing the informed consent form.
5. Patients who have experienced any degree of acute exacerbation of asthma or are experiencing an acute exacerbation of asthma within 4 weeks prior to screening.
6. Active infection or acute infection requiring systemic anti-infective therapy within 4 weeks prior to screening.
7. Presence of any severe and/or uncontrolled medical condition that, in the judgement of the investigator, affects the safety of the subject or interferes with the evaluation of the medication, including, but not limited to: severe neurological disease, history of serious mental disorders, major cardiovascular disease, diabetes mellitus that is poorly controlled on standardized therapy, presence of prolonged QTcF interval or cardiac arrhythmia, or immunodeficiency disorders.
8. Subjects with a history of liver disease or currently receiving treatment for liver disease during the screening period, including but not limited to acute and chronic hepatitis, cirrhosis or liver failure.
9. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg, and/or diastolic blood pressure ≥ 100 mmHg at screening or baseline).
10. Abnormal screening and baseline laboratory tests:

    1. White blood cell count < 3 × 109/L, or neutrophil count< 1.5 × 109/L, or platelet < 70 × 109/L, or hemoglobin < 90 g/L;
    2. Alanine aminotransferase (ALT) > 2 × ULN (upper limit of normal), or aspartate aminotransferase (AST) > 2 × ULN, or total bilirubin (TBIL) > 1.5 × ULN;
    3. Patients with moderate to severe renal insufficiency (eGFR < 60 ml/min/1.73m2, calculation of eGFR using the simplified MDRD equation);
    4. Screening positive for human immunodeficiency virus (HIV) or a positive syphilis antibody test, active hepatitis B virus infection (hepatitis B surface antigen positive and HBV-DNA load above the lower limit of detection) or active hepatitis C virus infection (HCV antibody positive and HCV-RNA load above the lower limit of detection).
11. Participation in a clinical trial of any other drug or medical device (treated with a drug or medical device in a clinical trial) within 3 months prior to screening.
12. Have undergone bronchial thermoplasty within 12 months prior to screening or plan to undergo this treatment during the study period.
13. Currently using or have used anti-interleukin-5 (IL-5) monoclonal antibody, anti-interleukin-4/13 (IL-4/13) monoclonal antibody, anti-interleukin-4 receptor (IL-4R) monoclonal antibody, anti-thymic stromal lymphopoietin (TSLP) monoclonal antibody, anti-IgE monoclonal antibody within 12 weeks prior to screening or within 5 half-lives of the drug, whichever is longer.
14. Patients who have previously received treatment with HSK31858 tablets or similar products of DPP1 inhibitors.
15. Patients who have used a strong inducer or inhibitor of CYP3A within 14 days or 5 half-lives prior to the first investigational product administration, whichever is longer.
16. Having received a drug that may cause hyperkeratosis of the skin (e.g., tumor necrosis factor alpha antagonist) within 4 weeks prior to screening.
17. Comorbidities associated with the development of non-hereditary palmoplantar keratoderma (e.g., myxedema, chronic lymphoedema).
18. Comorbid periodontal disease that, in the judgement of the investigator, has an impact on the study.
19. Currently smoking subjects or subjects who quit smoking within 6 months prior to the screening visit; previous smoking subjects with a smoking history >10 pack-year = packs per day × years of smoking (Note: 1 pack = 20 cigarettes, 10 pack-year = 1 pack/day × 10 years or 1/2 pack/day × 20 years).
20. History of drug use, or substance abuse within 2 years prior to screening.
21. Pregnant, or planning to become pregnant during the study, or breastfeeding.
22. Subjects judged by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-03-22 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
The annualized asthma exacerbation rate within 24 weeks | 24-week treatment period
  Total number of acute exacerbations of bronchial asthma occurring within 24 weeks of study dosing / actual length of follow-up within 24 weeks of dosing

SECONDARY OUTCOMES:
The annualized asthma exacerbation rate within 48 weeks | 48-week treatment period
  Total number of acute exacerbations of bronchial asthma occurring within 48 weeks of study dosing / actual length of follow-up within 48 weeks of dosing
Time to first acute exacerbation of bronchial asthma | 48-week treatment period
  Length of time from randomization to first acute exacerbation of bronchial asthma within 48 weeks of treatment
Change from Baseline in forced expiratory volume in 1 second (FEV1) | 48-week treatment period
  Change from baseline in pre-bronchodilator forced expiratory volume in 1 second (FEV1) at each clinical visit during the treatment period
Change from baseline in peak expiratory flow(PEF) | 48-week treatment period
  Change from baseline in peak expiratory flow (PEF) at each clinical visit during the treatment period
Change from baseline in Asthma Control Test (ACT) | 48-week treatment period
  Change from baseline in Asthma Control Test (ACT) score at each clinical visit during the treatment period.The ACT score is a questionnaire designed to assess the level of asthma control, including the impact of asthma on daily life, number of breathlessness episodes, asthma symptoms, use of rescue medication, and self-assessment of asthma control. The ACT score is a questionnaire designed to assess the level of asthma control, including the impact of asthma on daily life, number of breathlessness episodes, asthma symptoms, use of rescue medication, and self-assessment of asthma control.
Change from baseline in the 5-item Asthma Control Questionnaire (ACQ-5) | 48-week treatment period
  Change from baseline in the 5-item Asthma Control Questionnaire (ACQ-5) score at each clinical visit during the treatment period.5-item Asthma Control Questionnaire(ACQ-5) is a scoring scale used to assess asthma control in patients over the past week. It addresses asthma-related symptoms and consists of five items, each scored on a scale of 0 to 6, with higher scores indicating poorer control。Take the average score of 5 questions: <0.75 points indicate that asthma has been fully controlled; a score between 0.75 and 1.5 indicates that asthma is well controlled; and a score of >1.5 indicates that asthma is not controlled.
Change from baseline in 24-h sputum weight | 48-week treatment period
  Change from baseline in 24-h sputum weight at each clinical visit during the treatment period
The number of puffs of rescue medication used | 48-week treatment period
  The number of puffs of rescue medication used at each clinical visit during the treatment period
Change from baseline in Mini-Asthma Quality of Life Questionnaire (Mini-AQLQ) | 48-week treatment period
  Change from baseline in Mini-Asthma Quality of Life Questionnaire (Mini-AQLQ) scores after 12, 24, 36, and 48 weeks of treatment.The Mini-Asthma Quality of Life Questionnaire (Mini-AQLQ) is dedicated to assessing the quality of daily life in adults with asthma. The Asthma Quality of Life Questionnaire is a 7-point scale, with 1 indicating the worst and 7 the best. The sum of each item scores is the total score. The maximum total score is 105, with higher scores indicating better asthma control and lower scores indicating poorer quality of life.
The proportion of patients without acute exacerbation of bronchial asthma | 48-week treatment period
  The proportion of patients without acute exacerbation of bronchial asthma after 24 and 48 weeks of treatment
Patient Global Impression of Change (PGIC) | 48-week treatment period
  Patient Global Impression of Change (PGIC) after 24 and 48 weeks of treatment.The PGIC scale is an assessment of the overall change in the patient's condition since the start of the study and is rated on a 7-point scale: a score of 1 represents extreme improvement, 2 represents significant improvement, 3 represents slight improvement, 4 represents no improvement, 5 represents slight deterioration, 6 represents significant deterioration and 7 represents critical deterioration.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No